CLINICAL TRIAL: NCT04737304
Title: A First-in-Human, Double-Blind, Randomised, Vehicle Controlled Phase I/II Proof of Concept Study to Investigate the Safety, Tolerability, Pharmacokinetics and Efficacy of BEN2293 in Patients With Mild to Moderate Atopic Dermatitis
Brief Title: A First-in-Human PoC Study With BEN2293 in Patients With Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BenevolentAI Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BB-2293-101b
Record Dates: First submitted 2020-10-22; First posted 2021-02-03 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose Regimen Low Dose (Experimental): Low Dose Strength
  Interventions: Drug: BEN2293 (0.25% or 1.0% w/w) or matching placebo
- Dose Regimen High Dose (Experimental): High Dose Strength
  Interventions: Drug: BEN2293 (0.25% or 1.0% w/w) or matching placebo
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: BEN2293 (0.25% or 1.0% w/w) or matching placebo

INTERVENTIONS:
Drug: BEN2293 (0.25% or 1.0% w/w) or matching placebo — BEN2293 and placebo will be administered as a topical ointment. Both ointments contain the same excipients; placebo ointment has been manufactured in the same way except for the addition of 0.25% and 1.0% (w/w) BEN2293.
  Other Names: BEN2293

SUMMARY:
A randomised, adaptive design, double-blind, placebo-controlled, first-in-human, two-part study to investigate the safety, tolerability, PK and preliminary efficacy of multiple topical doses of BEN2293 in patients with mild to moderate AD.

DETAILED DESCRIPTION:
This Protocol will be adaptive and designed to enable knowledge gained from the previous cohort to be applied to subsequent cohorts. Changes made will be within the boundaries of the adaptive elements with clear control mechanisms and guidance for staying within these boundaries.

Part A is a randomised, double-blind, placebo-controlled, sequential group study to investigate ascending multiple topical doses of BEN2293 in patients with mild to moderate AD. Patients will participate in only one cohort.

Part B is a randomised, double-blind, placebo-controlled, parallel group study to investigate up to two dose regimens of topical doses of BEN2293 administered for a maximum of 28 days in patients with mild to moderate AD.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with mild to moderate AD (based on vIGA) free from other clinically significant illness or disease that may adversely affect the safety of the patient or the integrity of the study as determined by medical history, physical examination, safety laboratory and other assessments.
* History of AD for at least 6 months diagnosed by a dermatologist or GP.
* Previous or current successful treatment with topical corticosteroids.
* A vIGA score of 2 (mild) to 3 (moderate) at both Screening and Day -1 (Part A) and at Screening, Day-3 and Day 1 (Part B).

Exclusion Criteria:

* Atopic dermatitis of such severity that the patient could not comply with the demands of the study and/or the patient is not a suitable candidate for a placebo controlled study, as per Investigator's discretion.
* Any skin tattoo, scar, cuts, bruises, or other skin damage, including excessive UV exposure, at the possible IMP application sites.
* Patients who have AD lesions affecting >3% untreatable areas (face, scalp, genitals, palms of hands or soles of feet).
* Have concomitant skin disease or infection (e.g., acne, impetigo) or presence of skin comorbidities in the study area to be dosed that may interfere with study assessments.
* Patients who are excessively hirsute in areas of skin to be dosed with study ointment.
* Patients who are unwilling to stop hair removal by any means (including shaving, waxing or depilatory creams) to skin areas to be dosed with study ointment for 2 weeks prior to Day -1 and throughout the duration of the study.
* Clinically relevant history of abnormal physical or mental health interfering with the study as determined by medical history and physical examinations as judged by the Investigator (including [but not limited to], neurological, psychiatric, endocrine, cardiovascular, gastrointestinal, hepatic, or renal disorder).
* The patient has participated in a clinical study and has received a medication or a new chemical entity within 3 months prior to Day 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed by means of incidence of adverse events, incidence of adverse events at the local application site, mean vital signs, mean 12-lead ECG parameters and mean safety laboratory results. | Up to 28 days
  Parameters measured by prompted reporting of adverse events and scheduled safety assessments.

SECONDARY OUTCOMES:
PK-Cmax | Up to 28 days
  The investigation of the plasma PK of BEN2293 and metabolite BEN6403 following multiple topical doses to mild to moderate AD patients.
PK-Tmax | Up to 28 days
  The investigation of the plasma PK of BEN2293 and metabolite BEN6403 following multiple topical doses to mild to moderate AD patients.
PK-T1/2 | Up to 28 days
  The investigation of the plasma PK of BEN2293 and metabolite BEN6403 following multiple topical doses to mild to moderate AD patients.
PK-AUC | Up to 28 days
  The investigation of the plasma PK of BEN2293 and metabolite BEN6403 following multiple topical doses to mild to moderate AD patients.
PK- over a dosing interval (AUCт) | Up to 28 days
  The investigation of the plasma PK of BEN2293 and metabolite BEN6403 following multiple topical doses to mild to moderate AD patients.
PK - Accumulation ratio | Up to 28 days
  The investigation of the effect of BEN2293 on pruritus and Atopic Dermatitis in patients
Time to itch reduction | Up to 28 days
  The investigation of the effect of BEN2293 on pruritus and Atopic Dermatitis in patients with mild to moderate AD.
Fraction of patients achieving itch reduction | Up to 28 days
  The investigation of the effect of BEN2293 on pruritus and Atopic Dermatitis in patients with mild to moderate AD.
Change from baseline in the Numerical Rating Scale (NRS) for pruritus - Worst Itch over 24 hours | Up to 28 days
  The investigation of the effect of BEN2293 on pruritus and Atopic Dermatitis in patients with mild to moderate AD. Scale graded by 0 - no itch through to 10 - worst imaginable itch.
Change from baseline in the Numerical Rating Scale (NRS) for pruritus - Current Itch | Up to 28 days
  The investigation of the effect of BEN2293 on pruritus and Atopic Dermatitis in patients with mild to moderate AD. Scale graded by 0 - no itch through to 10 - worst imaginable itch.
Change from baseline in Eczema Area and Severity Index (EASI) score | Up to 28 days
  The investigation of the effect of BEN2293 on pruritus and Atopic Dermatitis in patients with mild to moderate AD. Index is graded 0 - none, absent, 1 - mild, 2 - moderate and 3 - severe.
Number of patients achieving improvement in Eczema Area and Severity Index (EASI) score | Up to 28 days
  The investigation of the effect of BEN2293 on pruritus and Atopic Dermatitis in patients with mild to moderate AD. Index is graded 0 - none, absent, 1 - mild, 2 - moderate and 3 - severe.
Change from baseline in BSA affected by AD in treated area(s) | Up to 28 days
  The investigation of the effect of BEN2293 on pruritus and Atopic Dermatitis in patients with mild to moderate AD.
Change from baseline in vIGA score | Up to 28 days
  The investigation of the effect of BEN2293 on pruritus and Atopic Dermatitis in patients with mild to moderate AD.
Change from baseline in Patient Oriented Eczema Measure (POEM) | Up to 28 days
  The investigation of the effect of BEN2293 on pruritus and Atopic Dermatitis in patients with mild to moderate AD. 7 questions based on skin condition graded between 0 - no days to 4 - everyday, with a total score of 28 being the worse.
Change from baseline in Dermatology Life Quality Index (DLQI) | Up to 28 days
  The investigation of the effect of BEN2293 on pruritus and Atopic Dermatitis in patients with mild to moderate AD. Index graded from 0 - not at all to 3 - very much. The higher the score, the more quality of life is impaired.
Change from baseline in EQ5D score | Up to 28 days
  The investigation of the effect of BEN2293 on pruritus and Atopic Dermatitis in patients with mild to moderate AD.
Change from baseline in Patient Reported Outcomes Measurement Information System (PROMIS) | Up to 28 days
  The investigation of the effect of BEN2293 on pruritus and Atopic Dermatitis in patients with mild to moderate AD. System has questions based on Itch - Scratching Behaviour, Itch - Mood and Sleep and Itch - Interference. questions are graded from 1 - never to 5 - almost always (worse score).
Change from baseline in Insomnia Severity Index (ISI) | Up to 28 days
  The investigation of the effect of BEN2293 on pruritus and Atopic Dermatitis in patients with mild to moderate AD. 7 questions based on quality of sleep, graded 0 - none to 4 - very severe. Total score of 28 being the worse.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Thompson, MBBS, Principal Investigator — MAC Clinical Research
Locations (1):
- MAC Clinical Research, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No